CLINICAL TRIAL: NCT06653309
Title: Interdisciplinary Pharmaceutical Analysis: Artificial Milk Effects on Neonates and Postnatal Women's Health
Brief Title: Interdisciplinary Pharmaceutical Analysis: Artificial Milk Effects on Children and Postnatal Women's Health
Acronym: Postnatal
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Basma Wageah Mohamed Mohamed Elrefay, Lecturer of obstetrics and gynaecology Nursing, Faculty of nursing- Delta University for Science and Technology, Egypt, Delta University for Science and Technology
Other Study IDs: Artificial Milk postnatal
Record Dates: First submitted 2024-10-14; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Breast Feeding
Keywords: Postnatal - Artificial Milk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- a natural breastfeeding and their corresponding postnatal women group: 100 a natural breastfeeding children, aged from 1 month to 1 year, and their corresponding postnatal women .
- artificial milk feeding group and their corresponding postnatal women group: 100 children, aged from 1 month to 1 year, and their corresponding postnatal women . children in this group is depending on artificial milk consumption .

SUMMARY:
Artificial milk, also known as infant formula, is a manufactured product designed to mimic the nutritional profile of human breast milk. Its biochemical composition is carefully crafted to provide a balanced mix of macronutrients, micronutrients, and other essential components that support the growth and development of infants . The primary macronutrients in artificial milk include carbohydrates, proteins, and fats, which are typically sourced from a combination of cow's milk, whey, and vegetable oils . Carbohydrates such as lactose and maltodextrins provide a quick source of energy, while proteins like whey protein and casein help to build and repair tissues. Fats like vegetable oils and medium-chain triglycerides (MCTs) provide essential fatty acids and help to support brain development .

In addition to these macronutrients, artificial milk also contains a range of micronutrients and other essential components that are important for infant health . These include vitamins like vitamin A, D, E, K, and C, as well as minerals like calcium, phosphorus, magnesium, and iron. Artificial milk may also contain added ingredients like DHA (docosahexaenoic acid) and ARA (arachidonic acid), which are important for brain and eye development . The exact composition of artificial milk can vary depending on the brand and type of formula, but most products are designed to meet the nutritional requirements established by organizations like the World Health Organization (WHO) and the American Academy of Pediatrics (AAP) . However, it is worth noting that the biochemical composition of artificial milk may not be identical to that of human breast milk, which is a complex mixture of nutrients and bioactive compounds that can provide unique benefits to infants .

DETAILED DESCRIPTION:
This study will employ a comparative observational design, involving a sample size of 200 children and their corresponding postnatal women. This design is a study in which the researcher is primary interested in describing relationships among variables, without seeking to establish a causal connection will utilize to conduct this study . The sample will be divided into two groups: a natural breastfeeding group and an artificial milk feeding group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 month and 1 year.
* Postnatal women who have given birth to a healthy neonate
* Postnatal women who are willing to participate in the study

Exclusion Criteria:

* • Children with major congenital anomalies or genetic disorders

  * Postnatal women with a history of breast surgery or trauma that may affect lactation
  * Postnatal women with a history of lactation insufficiency or nipple soreness

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 200 children, aged from 1 month to 1 year, and their corresponding postnatal women will provide sufficient power to detect statistically significant differences between the two groups, with a minimum of 100 participants in each group. Sample size was calculated using Open Epi I program at confidence interval 95% and power of 80%.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
increase global awareness about assessments of breast feeding and its difficulties | 3 months
  Nurses most often use a subjective "well/fair/poor" system to assess and document breastfeeding. LATCH is a breastfeeding charting system that provides a systematic method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. Each letter of the acronym LATCH denotes an area of assessment. "L" is for how well the infant latches onto the breast. "A" is for the amount of audible swallowing noted. "T" is for the mother's nipple type. "C" is for the mother's level of comfort. "H" is for the amount of help the mother needs to hold her infant to the breast. The system is visually represented in the same form as the Apgar scoring grid, and the numbers are handled in the same way. With the LA TCH system, the nurse can assess maternal and infant variables, define areas of needed intervention, and determine priorities in providing patient care and teaching

SECONDARY OUTCOMES:
raising awareness about the burden of depressive symptoms many women experience in postnatal women care | 3 months
  This tool was developed by Cox et al. (1996) (Cox et al., 1996). A standardized scale will be used to assess postnatal depression symptoms in postnatal women. The EPDS is a 10-item self-report scale assessing the common symptoms of depression.
  Scoring system Each item is scored on a 4-point scale (O-3), the minimum and maximum total score ranging from 0-30, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Basma Wageah Mohamed Mohamed Elrefay, Al Manşūrah, Al Dakahlya, Egypt